CLINICAL TRIAL: NCT06977711
Title: Phase Ib Clinical Trial of Loncastuximab and Roflumilast Added to R-CHOP (Lo-RR-CHOP) for Treatment Naïve High-Risk Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Loncastuximab and Roflumilast Added to R-CHOP (Lo-(Rituximab and Roflumilast) RR-CHOP) for Naïve High-Risk Diffuse Large B-cell Lymphoma (DLBCL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Adolfo Enrique Diaz Duque, Associate Professor/Clinical, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 24-0122; STUDY00001006 (Other: UT Health San Antonio)
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lymphoid neoplasms; Loncastuximab; Rituximab; Roflumilast; Lo-RR-CHOP; R-CHOP
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — loncastuximab tesirine; Roflumilast; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Prednisone

STUDY DESIGN:
Intervention Model Description: Phase I, single arm, open label clinical trial that
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Untreated High Risk DLBCL (Diffuse Large B-cell Lymphoma) (Experimental): Eligible subjects will receive 2 cycles of chemotherapy free therapy composed of Loncastuximab 0.15 mg/kg, Rituximab 375 mg/m2, and Roflumilast 500 ug po daily; followed by 6 cycles of chemoimmunotherapy with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) at standard of care (SOC) doses, and Roflumilast 500 ug po daily. Loncastuximab at a dose of 0.075 mg/kg will be added to other chemoimmunotherapy agents only for the first three (3) out of six (6) cycles
  Interventions: Drug: Loncastuximab; Drug: Roflumilast; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Loncastuximab — Intravenous (IV) administration 0.15 mg/kg day 1 cycles 1-2, and 0.075mg/kg day 1, cycles 3-5
Drug: Roflumilast — Oral administration of 500mcg days 1-21, cycles 1-8
Drug: Rituximab — IV administration of 375mg/m2 day 1, cycles 1-8
Drug: Cyclophosphamide — IV administration of 750mg/m2 day 1, cycles 3-8
Drug: Vincristine — IV administration 1.4mg/m2 (max 2mg) day 1, cycles 3-8
Drug: Doxorubicin — IV administration 50mg/m2 day 1, cycles 3-8
Drug: Prednisone — Oral administration 100mg/days 1-5, cycles 3-8

SUMMARY:
This study is developed by the investigator and is a, phase I, single arm, clinical trial that will enroll subjects with untreated diffuse large B-cell lymphoma (DLCBL) at high risk for poor outcome. The types of treatments given will be shared with participants.

The aims are:

1. To assess the safety and how well the participants tolerate the treatment
2. Assess the response of the tumor to treatment to estimate complete response
3. Assess the response of the tumor to treatment to estimate progression-free survival

DETAILED DESCRIPTION:
Exploratory analyses include cell free DNA (cfDNA). Each subject's disease will be biologically characterized at baseline.

Enrolled subjects will receive 2 cycles of chemotherapy free therapy composed of loncastuximab 0.15 mg/kg, rituximab 375 mg/m2, and roflumilast 500 ug po daily; followed by 6 cycles of chemoimmunotherapy with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) at standard of care (SOC) doses, in combination with loncastuximab and roflumilast 500 ug po daily. Loncastuximab at a dose of 0.075 mg/kg will be added to other chemoimmunotherapy agents only for the first three (3) out of six (6) cycles.

All subjects will have PET-CT at four time points during the trial: 1) screening, 2) cycle 3 (after the 2 initial chemotherapy free cycles of therapy), 3) cycle 6 (after 3 cycles of loncastuximab, roflumilast and R-CHOP), and 4) at end of therapy (EOT) after completing a total of eight cycles of treatment planned for the trial (two chemotherapy free and six of chemoimmunotherapy). All subjects will have cfDNA monitoring at three time points during the trial: 1) cycle 1 day 1 (baseline), 2) cycle 3 day 1 (after the 2 initial chemotherapy free cycles of therapy), and 3) at end of therapy (EOT) after completing a total of eight cycles of treatment planned for the trial (two chemotherapy free and six of chemoimmunotherapy). Responses will be evaluated by PET-CT as per Lugano response criteria1 and correlated with cfDNA analysis. Cycles are 21 days long.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older.
2. Pathologically proven diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS).

   - Patients with Diffuse large B-cell lymphoma/ high grade B-cell lymphoma with MYC (myelocytomatosis oncogene) and BCL2 (B-cell lymphoma 2) rearrangements are allowed.
3. No prior systemic therapy for lymphoma.
4. Subject has provided informed consent.
5. Subject is willing and able to comply with clinic visits and procedure outlined in the study protocol.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Life expectancy of ≥3 months.
8. Ann Arbor stage II-IV
9. National Comprehensive Cancer Network - International Prognostic Index (NCCN-IPI) risk score of ≥ 2
10. Measurable disease, meaning at least 1 lymph node or other lymphomatous lesion with a long axis of ≥1.5 cm by CT imaging, and at least one FDG-avid lesion by FDG-PET scan.
11. Left ventricular ejection fraction of at least 45% by either echocardiography or radionucleotide angiography.
12. Ability to swallow oral tablets without difficulty.
13. All subjects with preserved reproductive potential must agree to practice abstinence or employ contraceptive measures for the duration of treatment and for 10 months (if female) or 7 months (if male) following final dosing. All male subjects are considered to have reproductive potential.

    Female subjects of reproductive potential are those who:

    i) are not at least 50 years old and have no menses for 24 consecutive months; or ii) have not been rendered surgically sterile (having undergone hysterectomy and/or bilateral salpingo-oophorectomy).

    Female subjects of reproductive potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (hCG) within 7 days of first day of drug dosing.
14. Meet the following clinical laboratory requirements:

    * Creatinine clearance ≥30 ml/min by Cockcroft-Gault formula;
    * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (unless indirect bilirubin is elevated due to Gilbert's syndrome or hemolysis);
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤ 3 × ULN;
    * Platelet count ≥ 50,000/µL, with or without transfusion support;
    * Absolute Neutrophil Count (ANC) ≥ 1000/µL, with or without chronic granulocyte growth factor support;
    * Hemoglobin ≥8 g/dL, with or without transfusion support.

Exclusion Criteria:

1. Allergy or intolerance to roflumilast.
2. Allergy or intolerance to loncastuximab
3. Any active malignancy other than DLBCL
4. Current participation in another interventional clinical study
5. Prior allogeneic bone marrow transplant within 12 months of screening date.
6. Prior autologous stem cell transplant within 6 months of screening date.
7. Immunotherapy, chemotherapy, radiotherapy, or investigational therapy within 6 months prior to drug dosing.
8. Active central nervous system (CNS) involvement by lymphoma, including untreated symptomatic epidural disease.
9. Active uncontrolled infection.
10. Poorly controlled depressive symptoms and/ or currently under management for depression that is poorly controlled.
11. Significant disease or medical conditions, as assessed by the Investigator and Sponsor, that would substantially increase the risk benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV.
12. Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which subjects are not on active anti-cancer therapies and have had no evidence of active malignancy for at least 1 year.
13. History of major surgery within 3 weeks or minor surgery within 1 week of roflumilast administration. Major surgery includes, for example, any open or laparoscopic entry into a body cavity, or operative repair of fracture; minor surgery includes, for example, open surgical biopsy of palpable/superficial lymph node, or placement of vascular access device.
14. Other medical or psychiatric illnesses or organ dysfunction, which in the opinion of the investigator, would either compromise the subject's safety or interfere with the evaluation of the safety of the study agent.
15. Corrected QT interval (QTc) prolongation (defined as a QTc >450 ms for males and >470 ms for females -Fridericia's correction-) or other clinically significant ECG abnormalities as assessed by the investigator.
16. Baseline serum troponin above the upper limit of normal.
17. Baseline serum brain natriuretic peptide (BNP )above the age-adjusted upper limit of normal.
18. Baseline amylase above the upper limit of normal.
19. Subjects known to be HIV-positive must not have multi-drug resistant HIV infection, cluster of differentiation 4 (CD4) counts < 150/µl or other concurrent AIDS-defining conditions. Serologic screening for HIV is required within the 6 months prior to study enrollment.
20. Subjects positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C-virus ribonucleic acid (HCV RNA), unless both AST and ALT≤1.25 x ULN and there is no known history of chronic active hepatitis.

    Serologic screening for hepatitis B and C testing is required within the 6 months prior to study enrollment.
21. Subjects with moderate or severe liver impairment, as defined by a Child-Pugh class of B or C.
22. Women who are pregnant or breastfeeding.
23. Current use of any of the following medications: boceprevir, carbamazepine, ciprofloxacin, cobicistat, conivaptan, enzalutamide, fluvoxamine, itraconazole, ketoconazole, mitotane, phenytoin, posaconazole, rifampin, ritonavir, St. John's Wort, telaprevir, voriconazole, or zafirlukast.
24. Current use of non-nucleoside reverse transcriptase inhibitors (NNRTI) including efavirenz, rilpivirine, etravirine, delavirdine, nevirapine, and lersivirine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Estimation of number of adverse events | Baseline up to 8 cycles (up to 24 weeks)
  Estimation of adverse events (AE) and serious adverse events (SAE), graded according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

SECONDARY OUTCOMES:
Estimation of complete response | Baseline up to 8 cycles (up to 24 weeks)
  Estimation of complete response (CR) as defined by complete normalization of fluorodeoxyglucose positron emission tomography (FDG-PET) uptake (Deauville score of 1 to 3) of all target lesions
Estimation of progression-free survival (PFS) | Baseline up to 8 cycles (up to 24 weeks)
  Estimation of progression-free survival (PFS) defined as the time from the date of registration until the date of disease progression or death as a result of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo E Diaz Duque, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Ricardo Aguiar, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - University Hospital System, San Antonio, Texas
  - University of Texas Health Science Center San Antonio at the Cancer Therapy and Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
A description of study results will be provided at the end of the study. It will include a summary of overall entry status of all enrolled patients, and an account of all identified protocol violations. Patients who do not qualify for analysis, who die during the study, or who withdraw from the study before receiving treatment will be reported.
Supporting Information: Study Protocol, SAP
Time Frame: At study conclusion after data is analyzed and published in a peer review journal.